CLINICAL TRIAL: NCT06123416
Title: Emotion Regulation and Cancer Caregiving
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB-47800
Record Dates: First submitted 2019-01-17; First posted 2023-11-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Cancer; Healthy; Emotions
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Caregivers: Control participants will write about their daily and future tasks three times.
  Interventions: Behavioral: Expressive Writing
- Expressive Writing Caregivers: Experimental participants will write about their thoughts and feelings about an emotionally difficult event three times.
  Interventions: Behavioral: Expressive Writing

INTERVENTIONS:
Behavioral: Expressive Writing — Caregivers complete three 20-min writing sessions in which they write about an assigned topic - emotional or non-emotional.

SUMMARY:
The purpose of the study is to determine how the behaviors of cancer caregivers can impact patients.

ELIGIBILITY:
Inclusion Criteria:

All participants must:

* Be 21 years or older
* Have access to a computer with internet access

Patients must:

* Be women
* Have a diagnosis of breast cancer (non-recurrent)

Caregivers must be:

-The patient's caregiver (providing support to the patient)

Exclusion Criteria:

Participants must not be:

-Younger than 21 years

Patients must not:

* Be men
* Have a diagnosis other than breast cancer (non-recurrent)

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Nonrecurrent breast cancer patients and their caregivers (unpaid person who is close to the patient and provides emotional, medical and/or financial support).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire | Baseline through 3 months post-intervention
  Emotion regulation refers to the ways people influence which emotions they have, and how they experience and express these emotions. Participants will rate their habitual pursuit of pro-hedonic, contra-hedonic, pro-social, and impression management goals using the ERGS. The items will be rated on the same 7-point scale (1 = never; 7 = always).

CONTACTS AND LOCATIONS:
Overall Officials: Lameese Eldesouky, PhD, Principal Investigator — Stanford University; James Gross, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared it will only be shared upon request and will be de-identified.

REFERENCES:
- [Background] National Alliance for Caregiving. (2016). Cancer Caregiving in the U.S.: An Intense, Episodic, and Challenging Care Experience.
- [Background] Ryerson AB, Eheman CR, Altekruse SF, Ward JW, Jemal A, Sherman RL, Henley SJ, Holtzman D, Lake A, Noone AM, Anderson RN, Ma J, Ly KN, Cronin KA, Penberthy L, Kohler BA. Annual Report to the Nation on the Status of Cancer, 1975-2012, featuring the increasing incidence of liver cancer. Cancer. 2016 May 1;122(9):1312-37. doi: 10.1002/cncr.29936. Epub 2016 Mar 9. PMID 26959385
- [Background] Lwi SJ, Ford BQ, Casey JJ, Miller BL, Levenson RW. Poor caregiver mental health predicts mortality of patients with neurodegenerative disease. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):7319-7324. doi: 10.1073/pnas.1701597114. Epub 2017 Jun 27. PMID 28655841
- [Background] Kershaw, T., Northouse, L., Kritpracha, C., Schafenacker, A., & Mood, D. (2004). Coping strategies and quality of life in women with advanced breast cancer and their family caregivers. Psychology & Health, 19, 139-155.
- [Background] Appleton AA, Loucks EB, Buka SL, Kubzansky LD. Divergent associations of antecedent- and response-focused emotion regulation strategies with midlife cardiovascular disease risk. Ann Behav Med. 2014 Oct;48(2):246-55. doi: 10.1007/s12160-014-9600-4. PMID 24570218
- [Background] Gross, J. J. (1998). The emerging field of emotion regulation: An integrative review. Review of General Psychology, 2, 271-299.
- [Background] Gross, J. J. (2015). Emotion regulation: Current status and future prospects. Psychological Inquiry, 26, 1-26.
- [Background] Webb TL, Miles E, Sheeran P. Dealing with feeling: a meta-analysis of the effectiveness of strategies derived from the process model of emotion regulation. Psychol Bull. 2012 Jul;138(4):775-808. doi: 10.1037/a0027600. Epub 2012 May 14. PMID 22582737
- [Background] Srivastava S, Tamir M, McGonigal KM, John OP, Gross JJ. The social costs of emotional suppression: a prospective study of the transition to college. J Pers Soc Psychol. 2009 Apr;96(4):883-97. doi: 10.1037/a0014755. PMID 19309209
- [Background] Richards JM, Gross JJ. Emotion regulation and memory: the cognitive costs of keeping one's cool. J Pers Soc Psychol. 2000 Sep;79(3):410-24. doi: 10.1037//0022-3514.79.3.410. PMID 10981843
- [Background] Aldao A, Nolen-Hoeksema S, Schweizer S. Emotion-regulation strategies across psychopathology: A meta-analytic review. Clin Psychol Rev. 2010 Mar;30(2):217-37. doi: 10.1016/j.cpr.2009.11.004. Epub 2009 Nov 20. PMID 20015584
- [Background] Butler EA, Egloff B, Wilhelm FH, Smith NC, Erickson EA, Gross JJ. The social consequences of expressive suppression. Emotion. 2003 Mar;3(1):48-67. doi: 10.1037/1528-3542.3.1.48. PMID 12899316
- [Background] Pennebaker, J. W. (1997). Writing about emotional experiences as a therapeutic process. Psychological Science, 8, 162-166.
- [Background] Smyth JM. Written emotional expression: effect sizes, outcome types, and moderating variables. J Consult Clin Psychol. 1998 Feb;66(1):174-84. doi: 10.1037//0022-006x.66.1.174. PMID 9489272
- [Background] Zachariae R, O'Toole MS. The effect of expressive writing intervention on psychological and physical health outcomes in cancer patients--a systematic review and meta-analysis. Psychooncology. 2015 Nov;24(11):1349-59. doi: 10.1002/pon.3802. Epub 2015 Apr 14. PMID 25871981
- [Background] Ferrell B, Wittenberg E. A review of family caregiving intervention trials in oncology. CA Cancer J Clin. 2017 Jul 8;67(4):318-325. doi: 10.3322/caac.21396. Epub 2017 Mar 20. PMID 28319263
- [Background] Pennebaker JW. Putting stress into words: health, linguistic, and therapeutic implications. Behav Res Ther. 1993 Jul;31(6):539-48. doi: 10.1016/0005-7967(93)90105-4. PMID 8347112
- [Background] Lepore, S. J., & Smyth, J. (Eds.). (2003). The writing cure: How expressive writing influences health and well-being. Washington, DC: American Psychological Association.
- [Background] Pennebaker, J. W., & Graybeal, A. (2001). Patterns of natural language use: Disclosure, personality, and social integration. Current Directions in Psychological Science, 10, 90-93.
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Antoni MH, Lutgendorf SK, Cole SW, Dhabhar FS, Sephton SE, McDonald PG, Stefanek M, Sood AK. The influence of bio-behavioural factors on tumour biology: pathways and mechanisms. Nat Rev Cancer. 2006 Mar;6(3):240-8. doi: 10.1038/nrc1820. PMID 16498446
- [Background] Kim Y, Schulz R, Carver CS. Benefit-finding in the cancer caregiving experience. Psychosom Med. 2007 Apr;69(3):283-91. doi: 10.1097/PSY.0b013e3180417cf4. Epub 2007 Apr 9. PMID 17420443
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] Porter LS, Keefe FJ, Lipkus I, Hurwitz H. Ambivalence over emotional expression in patients with gastrointestinal cancer and their caregivers: associations with patient pain and quality of life. Pain. 2005 Oct;117(3):340-348. doi: 10.1016/j.pain.2005.06.021. PMID 16153771
- [Background] Pennebaker JW, Colder M, Sharp LK. Accelerating the coping process. J Pers Soc Psychol. 1990 Mar;58(3):528-537. doi: 10.1037//0022-3514.58.3.528. PMID 2324942
- [Background] Pennebaker JW, Kiecolt-Glaser JK, Glaser R. Disclosure of traumas and immune function: health implications for psychotherapy. J Consult Clin Psychol. 1988 Apr;56(2):239-45. doi: 10.1037//0022-006x.56.2.239. No abstract available. PMID 3372832
- [Background] Crawford J, Wilhelm K, Robins L, Proudfoot J. Writing for Health: Rationale and Protocol for a Randomized Controlled Trial of Internet-Based Benefit-Finding Writing for Adults With Type 1 or Type 2 Diabetes. JMIR Res Protoc. 2017 Mar 14;6(3):e42. doi: 10.2196/resprot.7151. PMID 28292741
- [Background] Kelley JE, Lumley MA, Leisen JC. Health effects of emotional disclosure in rheumatoid arthritis patients. Health Psychol. 1997 Jul;16(4):331-40. doi: 10.1037//0278-6133.16.4.331. PMID 9237085
- [Background] Riddle JP, Smith HE, Jones CJ. Does written emotional disclosure improve the psychological and physical health of caregivers? A systematic review and meta-analysis. Behav Res Ther. 2016 May;80:23-32. doi: 10.1016/j.brat.2016.03.004. Epub 2016 Mar 19. PMID 27017529
- [Derived] Eldesouky L, Gross JJ. Using expressive writing to improve cancer caregiver and patient health: A randomized controlled feasibility trial. Eur J Oncol Nurs. 2024 Jun;70:102578. doi: 10.1016/j.ejon.2024.102578. Epub 2024 Mar 21. PMID 38522170